CLINICAL TRIAL: NCT06581107
Title: Validate the Feasibility and Safety of the Robot System by Investgating the CT-fluoroscopy Guidance in Percutaneous Lung Cryablation Procedures of Participants With Lung Cancer
Brief Title: Validate the Safety and Feasibility of the CT-guided Interventional Robot in Percutaneous Lung Cryablation Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Wuhan United Imaging Surgical co., ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZRIR-002-24-06
Record Dates: First submitted 2024-08-29; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer; Thoracic Cancer
Keywords: Image-guided Biopsy; Robot-assisted procedures
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Singel arm (Experimental): CT-fluoroscopy guided robot-assisted percutaneous lung Cryoablation group
  Interventions: Procedure: CT-fluoroscopy guided master-slave intervetional robot-assisted lung Cryoablation

INTERVENTIONS:
Procedure: CT-fluoroscopy guided master-slave intervetional robot-assisted lung Cryoablation — During the procedure, the participants first undergo a CT scan. The radiologist plans the trajectories based on the registered preoperative CECT (contrast-enhanced computed tomography) and intraoperative CT. All participants then undergo navigation, localization, and establishment of cryoprobe trajectories using the interventional master-slave system. On the day of the procedure, the number of needle adjustments, number of cryoprobes used, puncture time, ablation time, and procedure time are recorded. The performance of the research device is evaluated by the radiologists. Postoperative complications of the participants are recorded 7±1 days postoperatively/on the day of discharge based on the postoperative CT scan (whichever comes first).

SUMMARY:
This study aims to investigate whether the interventional robot can be well and safely used for percutaneous lung cryoablation in patients with lung cancer. The robot allows radiologists to remotely control the needle insertion process under CT fluoroscopy guidance.

The main questions this study aims to answer are:

1. Whether the robot-assisted Cryoablation method can achieve complete the coverage of preoperatively planned ablation areas;
2. Whether the robot-assisted Cryoablation method can improve the success rate for radiologists to insert the needle into the target lesion area without additional needle adjustment;
3. Whether the robot-assisted Cryoablation method can reduce puncture time, ablation time and procedure time;
4. Whether the robot-assisted Cryoablation method can decrease the patient's complication occurrence rate;
5. Whether the robot-assisted Cryoablation method can obtain decent Evaluation of system performance.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of morbidity and mortality of malignant tumors.

The surgical resection of lung lobes is the standard treatment for stage I non-small cell lung cancer (NSCLC), with proven long-term cure rates and survival. However, more than 20% of patients are not eligible for surgical treatment due to comorbidities or poor underlying lung reserve.

With the development of minimally invasive interventional field, lung cancer cryoablation has also become an established tool for the treatment of early stage lung cancer and palliative treatment of advanced lung cancer in recent years.

However, the image-guidance cryoablation method still faces the following challenges:

1. Lack of real-time and accurate information during the needle insertion process, including puncture force, needle deformation, soft tissue deformation, and needle arrival position;
2. Multiple scans during the puncture are needed to determine whether the needle has successfully reached the target area, which leads to prolonged operation time, easily induces complications and increases the radiation dose to the physicians.
3. The accuracy of needle insertion is highly affected by the patient's respiration movement causing the multi-directional nonlinear displacement and deformation of tissues and organs (movement, rotation, etc.), resulting in the drift of the tumour position. Eventually, it is difficult for radiologists to reach the target position, resulting in insufficient ablation areas and increased probability of cancer recurrence.
4. The physiological trembling of the radiologist's hand will reduce the accuracy of puncture, and even lead to complications such as bleeding and pneumothorax
5. The procedure is highly dependent on the ability and experience of radiologists.

ELIGIBILITY:
Inclusion Criteria:

1. Participants suffering from lung cancer and judged by the investigator to be indicated for cryoablation procedures;
2. Participants voluntarily participate in this clinical study and sign the informed consent form;
3. Participants cannot undergo surgical treatment due to contraindications to surgical resection of lung cancer;
4. Participants can understand the study and cooperate with the study procedures, and are able to carry out follow-up observation as required.

Exclusion Criteria:

1. Participants have diffuse lesions in both lungs that cannot be improved by ablative therapy;
2. Participants suffer from extensive pleural metastases with massive pleural effusion;
3. Participants have tumors adjacent to the mediastinal blood vessels, contrast allergy, or inability to cooperate, which makes it difficult to choose the route of needle insertion;
4. Participants with lesions encircling blood vessels where ablation may lead to severe bleeding;
5. Participants with severely impaired lung function, with maximal ventilation <40%;
6. Participants with a low platelet count and severe coagulation abnormalities who cannot tolerate the procedure (anticoagulant therapy and/or anticoagulant medication should be discontinued for more than 1 week prior to ablation therapy);
7. Participants with poor general condition (multiple metastases throughout the body, severe infections, high fever), obvious malignant disease, severe insufficiency of vital organ function, severe anemia, and disorders of nutritional metabolism that cannot be improved in the short term;
8. Allergy to contrast media or anesthetics;
9. Pregnant or breastfeeding women, or those who plan to have children during the clinical study;
10. Participants with known addiction to drugs, alcohol, etc.;
11. Participants with psychiatric disorders who have no self-control and are unable to communicate clearly;
12. Participants who have participated in other drug, biologic, or medical device clinical studies without meeting the primary study endpoint timeframe prior to enrollment in this study;
13. Any other conditions that the investigator deems unsuitable for participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Technical success rate | The day of the procedure
  After the cryoablation procedure, the radiologists evaluate the consistency of the postoperative ablation area derived from the immediate postoperative thoracic CT scan with the size of the preoperative planning area. If consistent, it is defined as a technical success. The technical success rate is defined as the ratio of the number of participants with technical success to the total number of enrolled participants.

SECONDARY OUTCOMES:
The number of needle adjustments | The day of the procedure
  The number will be counted when the needle tip angle is altered or the needle is retracted during the procedure.
Number of cryoprobes used | The day of the procedure
  The number of cryoprobes used to complete cryoablation for a single target lesion during the cryoablation procedure.
Puncture time | The day of the procedure
  Time from when the needle tip enters the skin to the completion of the puncture.
Ablation time | The day of the procedure
  Time for the single lesion from when the cryoprobe arrives at the target to when the investigator judges the cryoablation is completed.
Procedure time | The day of the procedure
  Time from when the patient is positioned to the completion of the ablation procedure as judged by the investigator.
Evaluation of system performance | The day of the procedure
  Subjective evaluation from the radiologists regarding the commonly used functions, operation, stability, and convenience of the research device.
Compliations | 7±1 days postoperatively/on the day of discharge (whichever comes first).
  Complications including pneumothorax, hemoptysis, bleeding, and other rare complications.

CONTACTS AND LOCATIONS:
Overall Officials: Wenge Xing, Professor, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University, Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China